CLINICAL TRIAL: NCT02287142
Title: Evaluation of Supraclavicular, Suprascapular, and Interscalene Nerve Blocks for Outpatient Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, David Auyong, Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 14013
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Pain, Postoperative; Pain; Shoulder Joint; Pathologic Processes
MeSH Terms: conditions — Pain, Postoperative; Pain; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interscalene (Active Comparator): Single-shot Interscalene Nerve Block with ropivacaine 0.5%
  Interventions: Procedure: Brachial plexus nerve block
- Supraclavicular (Active Comparator): Single-shot Supraclavicular Nerve Block with ropivacaine 0.5%
  Interventions: Procedure: Brachial plexus nerve block
- Suprascapular (Active Comparator): Single-shot Suprascapular Nerve Block with ropivacaine 0.5%
  Interventions: Procedure: Brachial plexus nerve block

INTERVENTIONS:
Procedure: Brachial plexus nerve block — All arms of the study comparing the three different blocks are receiving the same single injection bolus of ropivacaine 0.5% prior to surgery. We will then record and compare pain scores in PACU and opioid requirement.

SUMMARY:
The aim of this study is to assess analgesic efficacy of a supraclavicular nerve block, suprascapular nerve block, or interscalene nerve block in a population undergoing shoulder arthroscopy with rotator cuff repair. The investigators hypothesize that subjects from all three arms will receive equal analgesia since these blocks are routinely performed to treat post-operative pain after shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral total shoulder arthroscopy for rotator cuff surgery ASA physical status I-III, >18 years old, Non-pregnant, Consent to participate in the study

Exclusion Criteria:

* Refusal to participate, < 18 years old, Chronic opioid use, Localized infection, Pregnancy or lactating, Pre-existing coagulopathy, Allergy to ultrasound gel or local anesthetics, Diaphragmatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain | Same day, 1 hour after arrival in the post-anesthesia care unit after surgery
  NRS Pain Scale

SECONDARY OUTCOMES:
Lung function | Same day, 1 hour after arrival in the post-anesthesia care unit after surgery
  Vital Capacity, Spirometry
Sensory and Motor Function | Same day, 1 hour after arrival in the post-anesthesia care unit after surgery
  Sensory Dermatome assessment C4 - C8 to touch; Motor assessment of grip and biceps with dynamometer
Diaphragmatic excursion | Same day, 1 hour after arrival in the post-anesthesia care unit after surgery
  Ultrasound measuring the diaphragm movement in centimeters (cm)

CONTACTS AND LOCATIONS:
Overall Officials: David Auyong, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States